CLINICAL TRIAL: NCT02936349
Title: Correlation of Graded Transthoracic Contrast Echocardiography With Chest CT Findings After Pulmonary Arteriovenous Malformation Embolization in Patients With Hereditary Hemorrhagic Telangiectasia, 2016
Brief Title: Graded TTCE for Post-Embolization PAVM Monitoring
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 825381
Record Dates: First submitted 2016-10-10; First posted 2016-10-18 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT)
Keywords: Hereditary Hemorrhagic Telangiectasia (HHT); Pulmonary Arteriovenous Malformation (PAVM); Transthoracic Contrast Echocardiogram (TTCE)
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Pulmonary Arteriovenous Fistulas

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Transthoracic Contrast Echocardiogram — A transthoracic contrast echocardiogram (TTCE) is a still or moving image of the internal parts of the heart using ultrasound following the injection of microbubble contrast (agitated saline) into a vein in the arm, which then travels to the heart.

SUMMARY:
Current HHT guidelines recommend CT scan to detect new or recurrent PAVMs after embolotherapy. Recent studies using transthoracic contrast echocardiography (TTCE) shunt grade for PAVM screening suggest that graded TTCE can accurately predict the size of PAVMs on chest CT and their amenability to embolization. This study's purpose is to evaluate whether TTCE shunt grade can also accurately predict PAVM size and amenability to treatment in patients who are post-embolization.

DETAILED DESCRIPTION:
Embolization is the standard of care for pulmonary arteriovenous malformations (PAVMs) in the Hereditary Hemorrhagic Telangiectasia (HHT) population. PAVMs are abnormal connections between the veins and arteries and result in right-to-left shunting of blood within the lungs. Successful embolization results in PAVM resolution and decreases the complications associated with right-to-left shunting. Current guidelines recommend follow-up with interval chest CT scan to determine treatment success and detect new or recurrent PAVMs after embolization. This results in significant radiation exposure to the relatively young HHT population. An alternative to chest CT is graded transthoracic contrast echocardiography (TTCE), which measures the amount of right-to-left shunting within the lung and assigns a grade based on this amount. TTCE has the advantage of being radiation free compared to chest CT. To date, graded TTCE has only been studied as a screening tool for PAVMs. These studies have shown that graded TTCE is highly sensitive in detecting PAVMs and is comparable to chest CT when screening for PAVMs. Results indicate that TTCE grade can accurately predict PAVM size on chest CT and predict whether PAVMs are amenable to embolization. However, no studies have compared graded TTCE and chest CT in patients who are post-embolization and it is therefore unknown whether graded TTCE can be used in patients who have undergone PAVM embolization. The current study seeks to correlate post-embolization TTCE grade with chest CT findings to determine whether TTCE can accurately predict PAVM size and amenability to treatment in the post-embolization population.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-89 years old
* Diagnosis of Hereditary Hemorrhagic Telangiectasia by the Curacao criteria
* Prior diagnosis of one or more PAVMs treated by embolotherapy
* Chest CT performed within the Penn system for surveillance of PAVMs after \ embolotherapy

Exclusion Criteria:

* Known PAVM recurrence on most recent chest CT with feeding artery size amenable to repeat embolotherapy
* Known history of intracardiac shunt
* Discovery of intracardiac shunt during transthoracic contrast echocardiography

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a diagnosis of Hereditary Hemorrhagic Telangiectasia and a follow-up chest CT scan for PAVM surveillance after embolotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Differences between TTCE shunt grade and the number of PAVMs present on most recent chest CT scan. | At the time of the echocardiogram (TTCE)
Differences between TTCE shunt grade and the size of PAVMs present on most recent | At the time of the echocardiogram (TTCE)

SECONDARY OUTCOMES:
Correlation between TTCE shunt grade to presence of PAVMs amenable to embolotherapy (feeding artery >2 mm) on most recent chest CT | 48 hours after echocardiogram (TTCE)

CONTACTS AND LOCATIONS:
Overall Officials: Scott O Trerotola, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DePietro DM, Curnes NR, Chittams J, Ferrari VA, Pyeritz RE, Trerotola SO. Postembolotherapy Pulmonary Arteriovenous Malformation Follow-Up: A Role for Graded Transthoracic Contrast Echocardiography Prior to High-Resolution Chest CT Scan. Chest. 2020 May;157(5):1278-1286. doi: 10.1016/j.chest.2019.11.023. Epub 2019 Nov 30. PMID 31794700